CLINICAL TRIAL: NCT05257161
Title: Independent Randomized Clinical Trial in Carotid Revascularization With MicroNet Covered Stent (CGuard) Comparing Early Neurological Outcomes With Distal EPS Versus Proximal EPS
Brief Title: Carotid Revascularization With MicroNet Covered Stent Comparing Early Neurological Outcomes With Distal Versus Proximal EPS
Acronym: SIBERIA-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Collaborators: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other); Chelyabinsk Regional Clinical Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIBERIA 2
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Patients With Aterosclerotic Carotid Stenosis; Symptomatic Patients (Stenosis > 50%); Asymptomatic Patients (Stenosis ≥80%)
Keywords: Carotid artery stenting. CGuard stent. Protection Device.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emboshield NAV6™ Embolic Protection System + CGuard™ (The CGuardTM Embolic Prevention System (EPS)) (Active Comparator): 183 Carotid stenting (Emboshield NAV6™ Embolic Protection System + CGuard™ (The CGuardTM Embolic Prevention System (EPS))
  Interventions: Device: Emboshield NAV6™
- MO.MA Proximal Cerebral Protection Device+ CGuard™ (The CGuardTM Embolic Prevention System (EPS) (Experimental): 183 Carotid stenting (MO.MA Proximal Cerebral Protection Device+ CGuard™ (The CGuardTM Embolic Prevention System (EPS))
  Interventions: Device: Mo.Ma™

INTERVENTIONS:
Device: Emboshield NAV6™ — Embolic Protection System for Carotid Artery Revascularization ( distal - filter) + stent CGuardTM™
  Other Names: Emboshield NAV6™ Embolic Protection System
  Arms: Emboshield NAV6™ Embolic Protection System + CGuard™ (The CGuardTM Embolic Prevention System (EPS))
Device: Mo.Ma™ — Embolic Protection System for Carotid Artery Revascularization ( proximal - occlusion) + stent CGuardTM™
  Other Names: Mo.Ma™ proximal cerebral protection device
  Arms: MO.MA Proximal Cerebral Protection Device+ CGuard™ (The CGuardTM Embolic Prevention System (EPS)

SUMMARY:
The SIBERIA study demonstrated a clear advantage of CGuard stent implantation over the existing classical stent when using a distal anti-embolic device. At the same time, there is no Level 1 evidence for a difference between the proximal and distal anti-embolic device for the CGuard stent.

ELIGIBILITY:
Inclusion Criteria

1. Consecutive patients 45-80 years old accepted for CAS following neurological consultation and qualification for the procedure according to center's routine practice.
2. More than 6-month life expectancy
3. Suitable clinical conditions for performing DW-MRI
4. Written Informed consent approved by the Ethics Committee
5. Subject agrees to all required follow-up procedures and visits

Exclusion Criteria:

1. Currently enrolled in another investigational device or drug study that has not completed the study or that clinically interferes with the current study endpoints
2. Recent surgical procedure within 30-days before or planned surgery within 30-days after the stenting procedure
3. Hepatic active disease (bilirubin> 35 mmol / l) or renal insufficiency (serum creatinine > 2.5 mg/dL or glomerular filtration rate <60 ml / min)
4. Recent evolving acute stroke within 30-days of study evaluation
5. Myocardial infarction within 72 hours prior to carotid stenting procedure (CPK-MB > 3 times normal)
6. Female patients of childbearing potential or known to be pregnant
7. Any known factor for potential stroke other than carotid stenosis, such as atrial fibrillation or atrial flutter (paroxysmal, permanent or persistent) or thrombophilia
8. Patient on VKA or new oral anticoagulants

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
determination of ischemic lesions | 24-48 hours
  Postprocedural acute ischemic lesions (MRI)

SECONDARY OUTCOMES:
MACCE | Intraoperatively, and within 48 hours.
  Death, stroke, and MI

CONTACTS AND LOCATIONS:
Locations (1):
- E. Meshalkin National Medical Research Center, Novosibirsk, Russia

REFERENCES:
- [Result] Montorsi P, Caputi L, Galli S, Ravagnani PM, Teruzzi G, Annoni A, Calligaris G, Fabbiocchi F, Trabattoni D, de Martini S, Grancini L, Pontone G, Andreini D, Troiano S, Restelli D, Bartorelli AL. Carotid Wallstent Versus Roadsaver Stent and Distal Versus Proximal Protection on Cerebral Microembolization During Carotid Artery Stenting. JACC Cardiovasc Interv. 2020 Feb 24;13(4):403-414. doi: 10.1016/j.jcin.2019.09.007. Epub 2020 Jan 29. PMID 32007460
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31855202/